CLINICAL TRIAL: NCT06206863
Title: Community-Based Physical Activity Across the Cancer Continuum
Brief Title: Community-Based Physical Activity Intervention for Underserved Cancer Survivors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: I 3414922; NCI-2023-10434 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 3414922 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2023-12-19; First posted 2024-01-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Hematopoietic and Lymphoid System Neoplasm; Malignant Solid Neoplasm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Supportive Care (virtual exercise classes) (Experimental): Participants participate in virtual exercise classes at least TIW over 20-60 minutes for 12 weeks. Participants are expected to work towards achieving the national physical activity exercise guidelines of 150 minutes of moderate intensity aerobic based physical activity and 2-3 strength training sessions each week.
  Interventions: Other: Exercise Intervention; Other: Questionnaire Administration

INTERVENTIONS:
Other: Exercise Intervention — Participate in virtual exercise classes
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial evaluates a community-based physical activity program for underserved cancer survivors. Cancer and its treatment significantly influence physical, psychosocial, and cognitive functioning. Historically, community sites (local and national) have not been staffed to offer support services such as physical, and occupational therapies (everyday life activities to promote health and well-being) or nutrition counselling, and do not offer a whole-person model of care. In this study, researchers have partnered with the YMCA to provide tailored home-based exercise programs for underserved cancer patients and survivors. Accessing exercise professionals may allow patients to prevent acute problems from becoming chronic, long-lasting physically weak impairments that directly influence patients' quality of life.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the feasibility and acceptability of a community-based 12-week physical activity intervention.

SECONDARY OBJECTIVE:

I. To assess the effectiveness of a virtual physical activity intervention by evaluating pre-post changes in quality of life (QoL).

EXPLORATORY OBJECTIVE (OPTIONAL):

I. To virtually assess changes in functional performance in a small subgroup.

OUTLINE:

Participants participate in virtual exercise classes at least three times a week (TIW) over 20-60 minutes for 12 weeks. Participants are expected to work towards achieving the national physical activity exercise guidelines of 150 minutes of moderate intensity aerobic based physical activity and 2-3 strength training sessions each week.

After completion of study intervention, patients are followed up at 1 week.

ELIGIBILITY:
Inclusion Criteria:

* Have had a previous cancer diagnosis OR are a caregiver for a patient who has had a previous cancer diagnosis
* Not in active treatment for cancer
* Over 18 years of age

Exclusion Criteria:

* Have uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, atrial fibrillation (AFIB), multiple myeloma, or psychiatric illness/social situations that would limit compliance with study requirements
* Have orthopedic or neuromuscular disorders or arthritis that preclude participation in exercise
* Are pregnant or nursing
* Are unwilling or unable to follow protocol requirements
* Have any condition which in the investigator's opinion deems the subject an unsuitable candidate to participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-08-20 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients referred to the intervention (Feasibility) | Up to 12 weeks
  At the provider level, feasibility will be defined as the proportion of patients that were referred to the intervention versus (vs.) the proportion of patients that enrolled in the study. Will estimate the referral rates with 95% confidence intervals obtained from generalized estimating equation (GEE) logistic regression models, accounting for the within provider clustering.
Proportion of patients that enrolled in the study (Feasibility) | Up to 12 weeks
  At the provider level, feasibility will be defined as the proportion of patients that were referred to the intervention vs. the proportion of patients that enrolled in the study.
Retention rate (Feasibility) | At the end of the 12-week intervention
  At the patient level, feasibility will be defined as the proportion of patients still on study. Will estimate with 95% confidence intervals obtained from GEE logistic regression models, accounting for the within provider clustering.
Adherence rate (Acceptability) | At post 12-weeks
  Adherence will be defined as the percentage of patients on study after 12-weeks who complete at least 70% of the intervention videos. Will estimate with 95% confidence intervals obtained from GEE logistic regression models, accounting for the within provider clustering.
Patient satisfaction (Acceptability) | Up to 12 weeks
  Acceptability will be determined by measuring adherence to the intervention and by measuring patient satisfaction. Patient satisfaction will be determined through pre-post intervention surveys. Will use the appropriate generalized linear model (ex. linear or logistic), as determined by the question type and accounting for the within provider clustering.

SECONDARY OUTCOMES:
Overall quality of life | Up to 12 weeks
  Will assess the changes in physical functioning, sustained physical activity, and quality of life using the European Organization for Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC QLQ-C30) score.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew D Ray, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States